CLINICAL TRIAL: NCT00420446
Title: The Effect of Daily Intakes of Dairy Products on Blood Pressure in Human Beings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: KA20060149
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2007-07-27 (Estimated); Status verified 2007-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

INTERVENTIONS:
Behavioral: Adjusted diet

SUMMARY:
The purpose of the project is to elucidate the effect on blood pressure by daily intake of dairy products. Previous studies have demonstrated a beneficial effect on blood pressure.

In total 90 subjects will be enrolled. For eight weeks, the participants will ingest one of two different dairy produces. Before, during and after the study period, the blood pressure is measured.

ELIGIBILITY:
Inclusion Criteria:

* Borderline hypertension

Exclusion Criteria:

* CVD, Diabetes, any kind of antihypertensive therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-01; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars T Jensen, M.D., Ph, Principal Investigator — Department of Clinical Physiology, Glostrup Hospital, DK-2600 Glostrup, Denmark; Hans Ibsen, M.D., D.M.Sc, Principal Investigator — Department of Internal Medicine M, Glostrup Hospital, DK-2600 Glostrup, Denmark
Locations (1):
- Department of clinical physiology, Glostrup Hospital, Glostrup Municipality, Denmark